CLINICAL TRIAL: NCT04203836
Title: A Phase 1, Randomised, Oral Dose Trial to Evaluate the Effect of Food on LEO 152020 in Healthy Adult Subjects
Brief Title: A Trial to Evaluate the Effect of Food on LEO 152020
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Collaborators: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: LP0190-1487
Record Dates: First submitted 2019-12-17; First posted 2019-12-18 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Healthy
Keywords: Healthy

STUDY DESIGN:
Intervention Model Description: Single dose, cross-over with food effect
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fed (Experimental): Single oral dose given after a full breakfast
  Interventions: Drug: LEO 152020 Tablet
- Fasting (Experimental): Single oral dose given in fasting state
  Interventions: Drug: LEO 152020 Tablet

INTERVENTIONS:
Drug: LEO 152020 Tablet — film-coated tablet

SUMMARY:
A phase 1 trial in healthy people to evaluate the food effect on LEO 152020 in an open-label design using film-coated tablets

DETAILED DESCRIPTION:
This trial will evaluate the pharmacokinetics and tolerability of 2 single doses of film-coated tablets in the morning after fasting or after a high-fat breakfast. The 2 doses will be separated by a washout period.

ELIGIBILITY:
Key inclusion Criteria:

* Body mass index (BMI) between 18.0-32.0 kg/m2 (both inclusive)
* In good health at screening and check-in as judged by the investigator based on medical history, physical examination, vital signs assessment, 12-lead ECG, and clinical laboratory evaluations.
* Pulse rate of 50 to 100 bpm at screening, or with minor deviations judged to be acceptable by the investigator
* Females of child bearing potential and male subjects whose partners are of child-bearing potential must also agree to use an additional effective method of contraception.

Key exclusion Criteria:

* Subjects who do not, or whose partners do not agree to use effective method(s) of contraception from the time of the first dose until 3 months (90 days) after the final dose.
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of any drug.
* History of any significant infectious disease within 2 weeks prior to drug administration as assessed by the investigator.
* Subjects who have received any medication within 14 days of the first dose administration, except for hormonal contraception.
* Subjects who are still participating in a clinical trial (e.g. attending follow-up visits) or who have participated in a clinical trial involving administration of an investigational drug (new chemical entity), or a marketed drug within the past 3 months prior to the first dose.
* ECG abnormalities at screening or check-in
* Heart rate of <50 or >100 beats per minute, unless the investigator judges the subject to be eligible for inclusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2020-12-12 (Actual); Study Completion 2020-12-12 (Actual)

PRIMARY OUTCOMES:
Cmax | pre-dose to 48 hours of each treatment period (Day 1 and Day 8)
  Maximum observed plasma concentration
AUC (0 to infinity) | pre-dose to 48 hours of each treatment period (Day 1 and Day 8)
  Area under the plasma concentration time curve (AUC) from time 0 extrapolated to infinity (AUC0 inf)

SECONDARY OUTCOMES:
Number of total adverse events (AEs) and number of subjects with AEs at each combination of treatment and period | Baseline to Day 10
  Number of AEs per subject at each combination of treatment and in total
Number of subjects with clinically relevant changes in vital signs (resting blood pressure) | Baseline to Day 10
  Clinically relevant changes in resting blood pressure (mmHq)
Number of subjects with clinically relevant changes in vital signs (pulse) | Baseline to Day 10
  Clinically relevant changes in pulse (beats per minute)
Number of subjects with clinically relevant changes in vital signs (oral body temperature) | Baseline to Day 10
  Clinically relevant changes in oral body temperature (fahrenheit/celsius)
Number of subjects with laboratory abnormalities in chemistry parameters | Baseline to Day 10
  Clinically relevant abnormalities in any chemistry laboratory parameters tested (standard units): Sodium, potassium, creatinine, creatine phosphokinase, urea nitrogen, calcium , alkaline phosphatase , aspartate aminotransferase , alanine aminotransferase , gamma glutamyl transferase , bilirubin, lactate dehydrogenase, cholesterol, triglycerides, glucose (fasting), albumin, protein, or tryptase
Number of subjects with laboratory abnormalities in haematology parameters | Baseline to Day 10
  Clinically relevant abnormalities in any haematology laboratory parameter tested (standard units): erythrocytes, hematocrit, hemoglobin, or white blood cells
Number of subjects with laboratory abnormalities in urinalysis parameters | Baseline to Day 10
  Clinically relevant laboratory abnormalities in any urinalysis parameters (standard units): protein, glucose, ketones, occult blood, leukocytes, or nitrite
Number of subjects with abnormal ECGs | Baseline to Day 10
  Abnormal ECGs (maximum QTcF interval of ≥450 msec, or maximum change from baseline of ≥60 msec)
AUC (0 to last) | pre-dose to 48 hours of each treatment period (Day 1 and Day 8)
  Area under the plasma concentration time curve (AUC) from time 0 extrapolated to infinity (AUC0 inf)
tmax | pre-dose to 48 hours of each treatment period (Day 1 and Day 8)
  Time to maximum plasma concentration
t 1/2 | pre-dose to 48 hours of each treatment period (Day 1 and Day 8)
  Terminal elimination half life

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (2):
- Leo Investigational Site, Dallas, Texas, United States
- LEO Pharma Investigational Site, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD can be made available to researchers in a closed environment for a specified period of time.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data is available to request after approval of the studied indication.
Access Criteria: Data-sharing is subject to approved scientifically sound research proposal and signed data-sharing agreement.
URL: http://leopharmatrials.com/for-professionals